CLINICAL TRIAL: NCT07104136
Title: Improvement of Adherence to Treatment Among COPD Patients in Primary Care by Physician-directed Intervention
Brief Title: Improving Adherence to COPD Treatments in Primary Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Clalit Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0195-24-COM1
Record Dates: First submitted 2025-07-16; First posted 2025-08-05 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Adherence to Care
Keywords: COPD; Primary care; Motivational interviewing; Inhalers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Randomization of primary care physicians to each group will be performed with stratification to the number of registered individual COPD patients for each physician. In addition, randomization will be performed with blocks of clinics from areas of similar sociodemographic characteristics.
Who Masked: Outcomes Assessor
Masking Description: Patients that will have their outcomes annalyzed will be unaware of group allocation or of the study considering data will be annalyzed retrospectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In the study, primary care physicians assigned to the intervention group will participate in a two-day seminar led by senior pulmonology specialists and family medicine specialists. The seminar will cover the following topic: Understanding COPD and current guidelines, inhaler technique and device selection, cardiovascular diseases in patients with COPD and possible interventions, motivational interview seminar, and two workshops for simulation and practice.
  The physicians will undergo a refresher workshop 3 months after entering the study, and visual and informative newsletter will be sent to them every 3 months.
  Interventions: Behavioral: COPD-care seminar
- Control (No Intervention): Primary care physicians that will be included without any intervention.

INTERVENTIONS:
Behavioral: COPD-care seminar — A two day seminar which will include:
  Lectures:
  Understanding COPD and Current Guidelines COPD pathophysiology. Review of the latest GOLD guidelines and treatment strategies Hands-on Session: Inhaler Technique and Device Selection Practical demonstration of different inhaler devices. Evaluating patient inspiratory effort and selecting suitable devices. Understanding advantages of each device and molecule. Cardiovascular diseases in COPD - real-world evidence, how to identify at-risk patients, and intervention.
  Motivational interview seminar- On line pre-course lectures about the theory behind motivational interview. Two workshops for simulation and practice of the technic through clinical cases with relevance to COPD patients including smoking cessation counseling techniques.
  Panel Discussion: Multidisciplinary Approach to COPD Management Involving respiratory specialists, physiotherapists, and primary care physicians.
  Discussion on referral practices and collaborative care.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to learn whether a special training program for primary care doctors can help improve treatment adherence and overall outcomes for people with chronic obstructive pulmonary disease (COPD).

The main questions it aims to answer are:

* Does the training program help patients with COPD take their medications more regularly?
* Does it reduce the number of COPD flare-ups (exacerbations)?
* Does it improve how well doctors follow current treatment guidelines for COPD?

In this study:

* Primary care doctors will be randomly assigned to either receive the training or continue their usual care without intervention.
* The training includes updated information about COPD, a workshop on inhaler use, and a course on motivational interviewing (a method to support behavior change)
* The care of their patients with COPD will be reviewed over 12 months to see if the program made a difference in medication use, flare-ups, and other outcomes.

DETAILED DESCRIPTION:
The investigators hypothesize that a primary care physician-directed intervention, consisting of a seminar with up-to-date professional guidance and motivational interviewing course, would result in patients' higher adherence to treatment, improved care, and fewer COPD exacerbations.

The study aims:

1. To evaluate the effect of specific COPD patient centric educational program for primary care physicians on adherence to recommended therapy.
2. To evaluate the effect of specific COPD patient centric educational program for primary care physicians on the number of moderate and severe COPD exacerbations.

This is a two-arm, parallel, randomized controlled trial conducted in a primary care setting, involving primary care physicians. All physicians will sign an informed consent form to participate.

The study will include two groups:

1. Intervention Group - Twenty primary care physicians will be recruited. After inclusion and signing an informed consent, all physicians will participate in a two-day seminar. The seminar will include: up-to-date professional guidance on COPD management, an inhalers workshop and a course of motivational interview. The physicians will undergo a refresher workshop 3 months after entering the study, and visual and informative newsletter will be sent to them every 3 months.
2. Control Group - Twenty primary care physicians, matched to the intervention group by sociodemographic area and number of COPD patients in past year.

The effect of the intervention will be assessed based on the outcomes of all COPD patients that visited one of the physicians in the intervention/control groups during the first 6 months after study initiation. These patients will be identified retrospectively from medical charts. Assessment of patient care and outcomes will be analyzed retrospectively, 18 months after study initiation (end of study), addressing each patient's first 12 months from first relevant clinic visit.

Randomization of primary care physicians to each group will be performed with stratification to the number of registered individual COPD patients for each physician. In addition, randomization will be performed with blocks of clinics from areas of similar sociodemographic characteristics.

COPD medication adherence rates vary by geographic location but are usually around 25-30%. Based on previous research, the investigators conservatively assume that our intervention will lead to an absolute 17% increase in adherence during the 12 months from first follow-up. Considering the above, to achieve an alpha of 0.05 and a power of 80%, there is a need for 127 patients in each group. Given that participating primary care physicians must have seen at least 18 individual COPD patients in the past year, and assuming a similar rate of visits during the follow-up period, along with a 15-20% loss-to-follow-up due to changes in the treating physician, the investigators estimate that 20 primary care physicians will be needed in each group.

ELIGIBILITY:
Inclusion Criteria:

* Primary care physicians
* Have at least 18 COPD patients in his unit as documented in medical records

Exclusion Criteria:

* Refusal to sign informed consent to participate in the study.
* Less than 1-year projection of employment in current clinic.
* Prior completion of a course in motivational interviewing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Adherence to COPD-related inhalers | From first patient visit after study initiation to 12 months after.
  Change in inhaler adherence from first clinic visit after trial initiation. Measured by the purchase of prescribed COPD inhalers and compared with the control group. The primary outcome will be assessed using the Proportion of Days Covered (PDC) method, calculated as the percentage of days a patient has medication available over the observation period. This outcome will be comapred between the intervention and control groups

SECONDARY OUTCOMES:
Change in adherence to inhaler therapy pre-post study | From first patient visit after study initiation to 12 months after.
  Change in inhaler adherence among COPD patients of primary care physicians in the 12 months prior and after inclusion, measured by the purchase of prescribed COPD medications and compared with the control group.
Non-inhaler medications adherence pre-post study | From first patient visit after study initiation to 12 months after.
  Non-inhaler medication adherence in the 12 months prior and after inclusion, measured by the purchase of prescribed COPD medications and compared with the control group.
Non-inhaler medication adherence | From first patient visit after study initiation to 12 months after.
  Non-inahler medication adherence from first clinic visit after study initiation, measured by the purchase of prescribed COPD medications and compared with the control group.
Annualized rate of moderate or severe COPD exacerbations | From first patient visit after study initiation to 12 months after.
  The difference in the annualized rate of moderate or severe COPD exacerbations between the intervention and control groups from first clinic visit after trial initiation. Moderate exacerbations are defined as those requiring treatment with systemic glucocorticoids, antibiotics, or both. Severe exacerbations are defined as those resulting in hospitalization or emergency medical care.
All-cause mortality | From first patient visit after study initiation to 12 months after.
  Incidence of all-cause mortality between the intervention and control
Cardiovascular events | From first patient visit after study initiation to 12 months after.
  The rate of patients with new cardiovascular events, including myocardial infarction, ischemic stroke, heart failure exacerbation leading to hospital, and cardiovascular-related mortality.
Guideline-based treatment | From first patient visit after study initiation to 12 months after.
  The percentage of patients at study end with inhaler therapy which meet the standard of care, as defined by the GOLD guidelines between the intervention and control groups
Physician knowledge on COPD | From first patient visit after study initiation to 12 months after.
  Evaluation of physicians knowledge about COPD and a questionnaire assessing whether, in the physician's opinion, the intervention has increased their knowledge and ability to treat patients with chronic obstructive pulmonary disease.

OTHER OUTCOMES:
New diagnoses of cardiovascular diseases - post hoc analysis | From first patient visit after study initiation to 12 months after.
  Rate of new diagnoses of cardiovascular diseases during the study period between the study groups, including diabetes, hypertension, hyperlipidemia, heart failure, coronary artery disease, peripheral vascular disease. Will be assessed by ICD codes.
Rate of guidelines-based cardiovascular treatment - post-hoc analysis | From first patient visit after study initiation to 12 months after.
  Rate of guidelines-based treatment for hypertension, diabetes, hyperlipidemia, and heart failure between the study groups. This outcome will be based on the ESC treatment guidelines.
Cardiovascular events - post-hoc analysis | From first patient visit after study initiation to 12 months after.
  Rate of cardiovascular events between the study groups, including heart failure exacerbation, myocardial infraction, and stroke.
Rate of cardio-pulmonary events - post-hoc analysis | From first patient visit after study initiation to 12 months after.
  The rate of cardio-pulmonary events, including COPD exacerbations, stroke, myocardial infraction, and heart failure exacerbations, between the study groups.
Time to first cardiovascular event - post-hoc analysis | From first patient visit after study initiation to 12 months after.
  Time to first cardiovascular event, including heart failure exacerbation, stroke, and myocardial infraction, between the study groups.
Control of cardiovascular risk - Post-hoc analysis | From first patient visit after study initiation to 12 months after.
  Rate of control of hypertension, diabetes, and hyperlipidemia, as assessed accoridng to the ESC guidelines between the groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Clalit health services, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
IPD might not be share due to limitations from the IRB committee

REFERENCES:
- [Background] Martinez FJ, Thomashow B, Sapir T, Simone L, Carter J, Han M. Does Evaluation and Management of COPD Follow Therapeutic Strategy Recommendations? Chronic Obstr Pulm Dis. 2021 Apr 27;8(2):230-242. doi: 10.15326/jcopdf.2020.0175. PMID 33610138